CLINICAL TRIAL: NCT06382857
Title: Effectiveness of a Microbiome-directed Food to Promote Programmatic and Sustained Nutritional Recovery Among Children With Uncomplicated Acute Malnutrition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: Epicentre, Niger (Unknown); National Nutrition Direction, Niger (Unknown); Ministry of Public Health and Social Affairs, Niger (Unknown); Regional Direction of Public Health, Maradi (Unknown)
Responsible Party: Principal Investigator, Sheila Isanaka, Associate Professor, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 823779-MDF Niger
Record Dates: First submitted 2024-04-16; First posted 2024-04-24 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Malnutrition, Child
Keywords: Malnutrition; SAM; MAM; Child; MDF; Microbiome
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition | interventions — milk-derived factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microbiome directed food (MDF) (Experimental): The MDF in this study was developed by the International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,B). This MDF is the lead icddr,B prototype that has demonstrated the strongest increase in biomarkers critical to growth, including growth hormone receptor and leptin, and re-establishment of the maturity of the microbiome among moderately malnourished children. Ingredients include chickpea flour, soy flour, peanut paste, green banana powder, sugar, oil, and micronutrients. The same MDF is provided for the treatment of SAM and MAM at modified doses.
  Interventions: Dietary Supplement: MDF
- Standard nutritional treatment (RUTF/RUSF) (Active Comparator): The standard RUTF used in this study for the treatment of SAM is Plumpy'Nut (Nutriset France). RUTF is a specialized therapeutic food that can be consumed without preparation and meets the nutritional requirements for the recovery of SAM. Ingredients include oil, peanut, skimmed milk powder, sugar and micronutrients. The standard RUSF used in this study is Plumpy'Sup (Nutriset France). RUSF is a lipid-based nutritional supplement with a high vitamin and mineral content, specifically designed for the treatment of MAM. Ingredients include oil, peanut, skimmed milk powder, sugar and micronutrients.
  Interventions: Dietary Supplement: RUTF; Dietary Supplement: RUSF

INTERVENTIONS:
Dietary Supplement: MDF — MDF will be provided to children on a weekly basis for children with SAM and bi-weekly basis for children with MAM at the health center until programmatic recovery but not thereafter.
  Arms: Microbiome directed food (MDF)
Dietary Supplement: RUTF — RUTF will be provided to all children on a weekly basis at the health center until programmatic recovery but not thereafter
  Other Names: Standard RUTF
  Arms: Standard nutritional treatment (RUTF/RUSF)
Dietary Supplement: RUSF — RUSF will be provided on a biweekly basis at the health center until programmatic recovery but not thereafter
  Other Names: Standard RUSF
  Arms: Standard nutritional treatment (RUTF/RUSF)

SUMMARY:
This study is an individually randomized controlled trial comparing microbiome-directed foods to standard nutritional therapy among children aged 6 to < 24 months with uncomplicated acute malnutrition in terms of programmatic recovery by 12 weeks from admission and sustained recovery at 24 weeks from admission.

ELIGIBILITY:
Inclusion Criteria:

* for children with Severe Acute Malnutrition (SAM): MUAC < 115 mm and/or WLZ < -3 and/or mild (+) or moderate (++) edema
* for children with Moderate Acute Malnutrition (MAM): 115 mm ≤ MUAC < 125 mm and/or -3 ≤ WHZ < -2
* Caregiver providing informed consent

Exclusion Criteria:

* Medical complications requiring inpatient treatment, as identified by the national protocol
* Not eating/lack of appetite (as informed by appetite test and investigator judgement)
* Re-admission into the program within 2 months of previous default
* for children with Severe Acute Malnutrition (SAM): Referral from inpatient care (therapeutic feeding center, TFC) or supplementary feeding program (SFP)
* for children with Moderate Acute Malnutrition (MAM): Referral from SAM treatment (TFC or OTP)
* Presence of congenital abnormality or underlying chronic disease that may affect growth or risk of infection
* Known contraindication/ hypersensitivity/allergy to study interventions (chickpea/soy flour, banana, peanut)
* Residence outside the study catchment area or in a non-fixed (e.g. nomadic) community

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7356 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Programmatic recovery by 12 weeks from admission | 12 weeks
  Defined as the proportion of SAM and MAM children achieving a WLZ ≥ -2 AND MUAC ≥ 125mm AND no edema during 2 consecutive visits
Sustained recovery at 24 weeks from admission | 24 weeks
  Proportion of recovered SAM and MAM children with WLZ ≥ -2 AND MUAC ≥ 125mm AND no edema

SECONDARY OUTCOMES:
Default | 12 weeks
  Defined as 2 consecutive missed scheduled program visits
Non-response | 12 weeks
  Defined as WLZ < -2 or MUAC < 125 mm during 2 consecutive visits, or for SAM children only: persistent edema at 12 weeks
Time to recovery | 12 weeks
  Measured as days from admission to programmatic recovery among recovered children
For MAM children: Deterioration to SAM | 24 weeks
  Weight-for-height z-score (WHZ) inferior to -3
Change in weight gain | From enrollment to 4, 8 and 12 weeks
  Change in g/kg/day
Change in weight-for-length Z (WLZ) | From enrollment to 4, 8 and 12 weeks
  Change in WLZ calculated using the 2006 WHO Growth Standards
Change in length-for-age Z (LAZ) | From enrollment to 4, 8 and 12 weeks
  Change in LAZ calculated using the 2006 WHO Growth Standards
Change in weight-for-age Z (WAZ) | From enrollment to 4, 8 and 12 weeks
  Change in WAZ calculated using the 2006 WHO Growth Standards
Change in MUAC | From enrollment to 4, 8 and 12 weeks
  Change in mm
Serious adverse events | 24 weeks
  Combined safety endpoint, including hospitalization and death
Hospitalization | 24 weeks
  Inpatient stay > 24h
Death | 24 weeks
  All-cause mortality
Motor, cognitive, language, social-emotional, and mental health skills | 24 weeks
  As measured by the Caregiver Reported Early Development Instrument (CREDI)
Cost effectiveness | 24 weeks
  As defined by the incremental cost per child recovered and per child sustained recovered
Dietary intake | 24 weeks
  As measured by 24h recall
Adherence | 12 weeks
  Defined as the sum of sachets returned used divided by the total number of sachets distributed
Microbiome profile at enrollment, week 4, program discharge, and study discharge | 24 weeks
  Defined as PCR-confirmed enteric viral, bacterial, and protozoan pathogens present
Plasma proteome profile at enrollment, week 4, program discharge, and study discharge | 24 weeks
  Defined as circulating plasma proteins (IGFBP-2, thrombospondin-5, granulysin, GDF-15, and MMP-8)
Environmental enteric dysfunction at enrollment, program discharge, and study discharge | 24 weeks
  Measured by anti-LPS IgA and IgG; anti-flagellin IgA and IgG; sCD14; I-FABP; myeloperoxidase (MPO); and calprotectin
Change of fat mass and fat-free mass at program discharge and study discharge | 24 weeks
  Measured by deuterium dilution
Micronutrient status at enrollment, program discharge and study discharge | 24 weeks
  Defined as ferritin; soluble transferrin binding protein; alpha-tocopherol; retinol; folate; and vitamin B12
Immuno-sufficiency at week 2, week 4, program discharge, week 12 and study discharge (SAM only) | 24 weeks
  As defined by T-cell receptor excision circles (TRECs) and kappa-receptor excision circles (KRECs)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Grais, PhD, Study Chair — Epicentre
Locations (1):
- Epicentre Niger, Maradi, Niger

IPD SHARING:
Plan to Share IPD: No